CLINICAL TRIAL: NCT01717755
Title: Basilar Artery International Cooperation Study
Acronym: BASICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erik van der Hoeven (Other)
Collaborators: BASICS Study Group (Unknown)
Responsible Party: Sponsor-Investigator, Erik van der Hoeven, E.J.R.J. van der Hoeven, MD, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL33550.100.10; NHS2010B151 (Other Grant/Funding Number: Dutch Heart Foundation); 2010-023507-95 (EudraCT Number)
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Basilar Artery Thrombosis; Basilar Artery Embolism; Stroke of Basilar Artery; Stroke; Cerebrovascular Disorders; Basilar Artery Occlusion
Keywords: basilar; stroke; mechanical; thrombolysis; intra-arterial; trombectomy
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best medical management. (No Intervention): Best medical management consists of the standard of care of patients with acute ischemic stroke according to existing local protocols and guidelines, and may include IV thrombolysis.
  If treated with IVT as part of BMM, IVT should be started within 4.5 hours of estimated time of BAO.
- Additional intra-arterial treatment. (Experimental): Best medical management followed by intra-arterial treatment and best medical management
  Interventions: Other: Intra-arterial treatment

INTERVENTIONS:
Other: Intra-arterial treatment — IA therapy has to be initiated within 6 hours of estimated time of basilar artery occlusion. If an appropriate thrombus or residual stenosis is identified, the choice of IA strategy wil be made by the treating neurointerventionalist. Choice of therapy depends on local approval and experience. If IA thrombolysis is the chosen strategy, a maximum of 22 mg of IA rt-PA or 1.500.000 Units of Urokinase may be given. Stenting is allowed in the presence of a high-grade vertebral artery stenosis or occlusion hampering adequate endovascular access to the basilar artery and in case of a residual high-grade basilar artery stenosis. The use of any other treatment strategy depends on local approval and experience, and is only allowed after prior approval of the steering committee.
  Arms: Additional intra-arterial treatment.

SUMMARY:
Rationale: Recently our study group reported the results of the Basilar Artery International Cooperation Study (BASICS), a prospective registry of patients with an acute symptomatic basilar artery occlusion (BAO). Our observations in the BASICS registry underscore that we continue to lack a proven treatment modality for patients with an acute BAO and that current clinical practice varies widely. Furthermore, the often-held assumption that intra-arterial thrombolysis (IAT) is superior to intravenous thrombolysis (IVT) in patients with an acute symptomatic BAO is challenged by our data. The BASICS registry was observational and has all the limitations of a non-randomised study. Interpretation of results is hampered by the lack of a standard treatment protocol for all patients who entered the study.

Objective: Evaluate the efficacy and safety of IAT in addition to best medical management (BMM) in patients with basilar artery occlusion.

Study design: Randomised, multi-centre, open label, controlled phase III, treatment trial.

Study population: Patients, aged 18 years and older, with CTA or MRA confirmed basilar occlusion.

Intervention: Patients will be randomised between BMM with additional IAT versus BMM alone. IAT has to be initiated within 6 hours from estimated time of BAO. If treated with as part of BMM, IVT should be started within 4.5 hours of estimated time of BAO.

Main study parameters/endpoints: Favorable outcome at day 90 defined as a modified Rankin Score (mRS - functional scale) of 0-3.

ELIGIBILITY:
Inclusion criteria

* Symptoms and signs compatible with ischemia in the basilar artery territory.
* Basilar artery occlusion (BAO) confirmed by CTA or MRA.
* Age 18 years or older (i.e., candidates must have had their 18th birthday).
* If IVT is considered as part of best medical management, IVT should be started within 4.5 hours of estimated time of BAO. (Estimated time of BAO is defined as time of onset of acute symptoms leading to clinical diagnosis of BAO or if not known last time patient was seen normal prior to onset of these symptoms).
* Initiation of IAT should be feasible within 6 hours of estimated time of BAO.

Exclusion criteria

* Pre-existing dependency with mRankin ≥3.
* Females of childbearing potential who are known to be pregnant and/or lactating or who have positive pregnancy tests on admission.
* Patients who require hemodialysis or peritoneal dialysis.
* Other serious, advanced, or terminal illness.
* Any other condition that the investigator feels would pose a significant hazard to the patient if thrombolytic therapy is initiated.
* Current participation in another research drug treatment protocol (patient cannot start another experimental agent until after 90 days).
* Informed consent is not or cannot be obtained.

Imaging exclusion criteria

* High-density lesion consistent with hemorrhage of any degree.
* Significant cerebellar mass effect or acute hydrocephalus.
* Bilateral extended brainstem ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2011-10; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Favourable outcome | day 90
  Favourable outcome at day 90 defined as a modified Rankin Score (mRS - functional scale) of 0-3.

SECONDARY OUTCOMES:
Excellent outcome | day 90
  Excellent outcome at day 90 defined as a modified Rankin Score (mRS - functional scale) of 0-2.
Modified Rankin Score | day 90
  Modified Rankin Score - not dichotomized.
NIHSS | pre IVT, pre randomization, 24h post treatment
  National Institutes of Health Stroke Scale (NIHSS - acute assessment scale) at timepoints:
  * directly pre intravenous thrombolysis
  * directly pre randomization (post intravenous thrombolysis)
  * at 24 hours +- 6 hours post treatment.
EQ-5D | day 90 and 12 months
  EQ-5D (quality of life) at day 90 and at 12 months.

OTHER OUTCOMES:
Recanalization | 24 hours ± 6 hours
  Recanalization at 24 hours ± 6 hours, by CT angiography.
Volume of cerebral infarction | 24 hours ± 6 hours
  Volume of cerebral infarction on NCCT and CTA source images.
SICH | 24 hours ± 6 hours.
  Symptomatic intracranial hemorrhage at 24 hours CT imaging ± 6 hours.
Mortality | 90 days
  Mortality at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: W J Schonewille, MD, Principal Investigator — St. Antonius Hospital
Locations (27):
- Brazil (2):
  - Fortaleza General Hospital, Fortaleza
  - Hospital das Clinicas de Ribeirao Preto, Ribeirão Preto
- Germany (5):
  - Klinikum Augsburg, Augsburg
  - Berlin Charite Hospital, Berlin
  - Dresden University Hospital, Dresden
  - University Medical Center Mannheim, Mannheim
  - Oberschwabenklinik, Ravensburg
- Italy (6):
  - Bergamo Hospital, Bergamo
  - Genova Hospital, Genoa
  - University Hospital Modena, Modena
  - Santa Corona Hospital, Pietra Ligure
  - Roma Umberto I, Rome
  - Varese Hospital, Varese
- Netherlands (11):
  - Rijnstate, Arnhem, Gelderland
  - Academic Hospital Maastricht, Maastricht, Limburg
  - St. Elisabeth Hospital, Tilburg, North Brabant
  - Academic Medical Center, Amsterdam, North Holland
  - MCH Westeinde, The Hague, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - University Medical Center Groningen, Groningen
  - Leiden University Hospital, Leiden
  - Erasmus Medical Center, Rotterdam
  - Haga Hospital, The Hague
  - Universitary Medical Center Utrecht, Utrecht
- Norway (2):
  - University Hospital North Norway, Tromsø
  - St. Olavs Hospital Trondheim, Trondheim
- University Hospital of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Schonewille WJ, Wijman CA, Michel P, Rueckert CM, Weimar C, Mattle HP, Engelter ST, Tanne D, Muir KW, Molina CA, Thijs V, Audebert H, Pfefferkorn T, Szabo K, Lindsberg PJ, de Freitas G, Kappelle LJ, Algra A; BASICS study group. Treatment and outcomes of acute basilar artery occlusion in the Basilar Artery International Cooperation Study (BASICS): a prospective registry study. Lancet Neurol. 2009 Aug;8(8):724-30. doi: 10.1016/S1474-4422(09)70173-5. Epub 2009 Jul 3. PMID 19577962
- [Background] Greving JP, Schonewille WJ, Wijman CA, Michel P, Kappelle LJ, Algra A; BASICS Study Group. Predicting outcome after acute basilar artery occlusion based on admission characteristics. Neurology. 2012 Apr 3;78(14):1058-63. doi: 10.1212/WNL.0b013e31824e8f40. Epub 2012 Mar 21. PMID 22442438
- [Background] Vergouwen MD, Compter A, Tanne D, Engelter ST, Audebert H, Thijs V, de Freitas G, Algra A, Jaap Kappelle L, Schonewille WJ. Outcomes of basilar artery occlusion in patients aged 75 years or older in the Basilar Artery International Cooperation Study. J Neurol. 2012 Nov;259(11):2341-6. doi: 10.1007/s00415-012-6498-2. Epub 2012 Apr 18. PMID 22527236
- [Background] Puetz V, Khomenko A, Hill MD, Dzialowski I, Michel P, Weimar C, Wijman CA, Mattle HP, Engelter ST, Muir KW, Pfefferkorn T, Tanne D, Szabo K, Kappelle LJ, Algra A, von Kummer R, Demchuk AM, Schonewille WJ; Basilar Artery International Cooperation Study (BASICS) Group. Extent of hypoattenuation on CT angiography source images in basilar artery occlusion: prognostic value in the Basilar Artery International Cooperation Study. Stroke. 2011 Dec;42(12):3454-9. doi: 10.1161/STROKEAHA.111.622175. Epub 2011 Sep 29. PMID 21960577
- [Background] Arnold M, Fischer U, Compter A, Gralla J, Findling O, Mattle HP, Kappelle LJ, Tanne D, Algra A, Schonewille WJ; BASICS Study Group. Acute basilar artery occlusion in the Basilar Artery International Cooperation Study: does gender matter? Stroke. 2010 Nov;41(11):2693-6. doi: 10.1161/STROKEAHA.110.594036. Epub 2010 Oct 14. PMID 20947845
- [Background] Schonewille WJ, Wijman CA, Michel P, Algra A, Kappelle LJ; BASICS Study Group. The basilar artery international cooperation study (BASICS). Int J Stroke. 2007 Aug;2(3):220-3. doi: 10.1111/j.1747-4949.2007.00145.x. PMID 18705948
- [Background] Schonewille W, Wijman C, Michel P; BASICS investigators. Treatment and clinical outcome in patients with basilar artery occlusion. Stroke. 2006 Sep;37(9):2206; author reply 2207. doi: 10.1161/01.STR.0000237127.84408.c0. Epub 2006 Aug 10. No abstract available. PMID 16902170
- [Background] Vergouwen MD, Algra A, Pfefferkorn T, Weimar C, Rueckert CM, Thijs V, Kappelle LJ, Schonewille WJ; Basilar Artery International Cooperation Study (BASICS) Study Group. Time is brain(stem) in basilar artery occlusion. Stroke. 2012 Nov;43(11):3003-6. doi: 10.1161/STROKEAHA.112.666867. Epub 2012 Sep 18. PMID 22989501
- [Derived] Roaldsen MB, Jusufovic M, Berge E, Lindekleiv H. Endovascular thrombectomy and intra-arterial interventions for acute ischaemic stroke. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD007574. doi: 10.1002/14651858.CD007574.pub3. PMID 34125952
- [Derived] Langezaal LCM, van der Hoeven EJRJ, Mont'Alverne FJA, de Carvalho JJF, Lima FO, Dippel DWJ, van der Lugt A, Lo RTH, Boiten J, Lycklama A Nijeholt GJ, Staals J, van Zwam WH, Nederkoorn PJ, Majoie CBLM, Gerber JC, Mazighi M, Piotin M, Zini A, Vallone S, Hofmeijer J, Martins SO, Nolte CH, Szabo K, Dias FA, Abud DG, Wermer MJH, Remmers MJM, Schneider H, Rueckert CM, de Laat KF, Yoo AJ, van Doormaal PJ, van Es ACGM, Emmer BJ, Michel P, Puetz V, Audebert HJ, Pontes-Neto OM, Vos JA, Kappelle LJ, Algra A, Schonewille WJ; BASICS Study Group. Endovascular Therapy for Stroke Due to Basilar-Artery Occlusion. N Engl J Med. 2021 May 20;384(20):1910-1920. doi: 10.1056/NEJMoa2030297. PMID 34010530
- [Derived] van der Hoeven EJ, Schonewille WJ, Vos JA, Algra A, Audebert HJ, Berge E, Ciccone A, Mazighi M, Michel P, Muir KW, Obach V, Puetz V, Wijman CA, Zini A, Kappelle JL; BASICS Study Group. The Basilar Artery International Cooperation Study (BASICS): study protocol for a randomised controlled trial. Trials. 2013 Jul 8;14:200. doi: 10.1186/1745-6215-14-200. PMID 23835026